CLINICAL TRIAL: NCT06855420
Title: Investigating the Efficacy of Foot Sole Vibration on Balance and Physical Activity in People with Diabetic Peripheral Neuropathy.
Brief Title: Smart Insoles for Improving Sensation, Balance and Mobility in People with Diabetic Peripheral Neuropathy.
Acronym: Pathfeel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walk With Path (Industry)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 46201
Record Dates: First submitted 2024-11-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathies; Unsteadiness
Keywords: smart wearable device; vibration; insoles; gait; peripheral sensation; balance
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibration (Active Comparator): Insoles with vibration
  Interventions: Device: Vibration on
- No Vibration (Placebo Comparator): Insoles without vibration
  Interventions: Device: Vibration off

INTERVENTIONS:
Device: Vibration on — Sole vibration will be applied by a vibrating insole system for 10 days. Participants will wear the device for at least 4 hours per day.
  Arms: Vibration
Device: Vibration off — Participants will wear the device with vibration turned off for at least 4 hours per day during 10 days of intervention.
  Arms: No Vibration

SUMMARY:
The long-term effects of vibrating insoles on improving gait, balance and peripheral sensation in people with diabetic peripheral neuropathy remain unknown. The Pathfeel Clinical Trial will investigate the efficacy of vibratory insoles worn for ten days for enhancing sensory perception, gait quality, balance and physical activity in people with mild to severe diabetic neuropathy. The primary outcome will be changes in gait speed and postural and dynamic balance.

DETAILED DESCRIPTION:
The Path Feel Clinical Trial will investigate the efficacy of foot sole vibration applied for 10 days during daily life for improving peripheral sensation, balance and mobility in people with diabetic peripheral neuropathy.

Twenty-two people with mild to severe diabetic neuropathy will perform a prospective comparison where they wear an insole system over the course of two interventional periods of 10 days each in a randomised, cross-over design, during which there will be a period where the device provides vibrational stimuli, vs a control condition where the device is worn, but provides no stimuli. Any changes in activity levels, peripheral sensation, quality of life and balance control will be compared between each condition to determine the longer-term effects of foot sole vibration.

Each participant will undertake four study visits with periods of device use between them. Participants will complete a set of questionnaires that will assess quality of life (NeuroQoL) and fear of falling (FES-I). Measurements of the level of peripheral neuropathy will be taken at both feet using non-invasive methods, including a neurothesiometer (i.e., Vibration Perception Threshold) and a composite score (i.e., modified Neuropathy Disability Score). Gait, postural and dynamic balance during daily activities, including walking, stair walking will be assessed through a combination of 3D Motion Capture system and force platforms. Changes in physical activity will be quantified by accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes type 1 or 2
* ≥1 palpable foot pulses
* Presence of mild to moderate diabetic peripheral neuropathy defined by a vibration perception threshold ≥15 Volts and/or mNDS score ≥3.
* Aged ≥ 18 years
* Ability to walk unaided for 30 steps
* Able to understand the study requirements
* Ability to check their feet regularly (or have another person check).
* Able to read the study documents
* Fit shoe size EU 36-47.5 / UK 3.5-13.

Exclusion Criteria:

• Active foot ulcer

* Lower limb amputation (anything more than amputation of two lesser toes)
* Presence of Charcot deformity
* Dementia or other cognitive impairment
* Significant cardiopulmonary or other systemic disease limiting the patient's ability to walk 30 steps.
* Person's with bodyweight greater than 130kg (due to insole device limitations)
* Presence of implantable neurostimulators
* Presence of a pacemaker.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Postural Balance | Measurements were taken at four time points: at baseline, after 10 days of the first vibratory intervention, after a 10-day washout period, and at the end of the 10-day second vibratory intervention.
  Centre-of-pressure velocity will be assessed using a force platform.
Gait speed during walking | Measurements were taken at four time points: at baseline, after 10 days of the first vibratory intervention, after a 10-day washout period, and at the end of the 10-day second vibratory intervention.
  Gait speed during level and stair walking will be assessed by 3D Motion Capture system.

SECONDARY OUTCOMES:
Peripheral Sensation | Measurements were taken at four time points: at baseline, after 10 days of the first vibratory intervention, after a 10-day washout period, and at the end of the 10-day second vibratory intervention.
  Vibration perception threshold (VPT) at the hallux will be measured bilaterally by a neurothesiometer.
Peripheral Sensation 2 | Measurements were taken at four time points: at baseline, after 10 days of the first vibratory intervention, after a 10-day washout period, and at the end of the 10-day second vibratory intervention.
  Large and small sensory nerve function will be assessed using the modified Neuropathy Disability Score (mNDS), a composite scoring tool ranging from 0 to 10 points. Higher scores indicate a greater decline in sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Neil D. Reeves, PhD, Professor, Principal Investigator — Lancaster University
Locations (1):
- Manchester Metropolitan University, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Orlando G, Brown S, Jude E, Bowling FL, Boulton AJM, Reeves ND. Acute Effects of Vibrating Insoles on Dynamic Balance and Gait Quality in Individuals With Diabetic Peripheral Neuropathy: A Randomized Crossover Study. Diabetes Care. 2024 Jun 1;47(6):1004-1011. doi: 10.2337/dc23-1858. PMID 38536962